CLINICAL TRIAL: NCT06969937
Title: Phase II, Randomised, Placebo-controlled, Double Blind, Parallel Group, Single Centre Study Investigating Ketamine and Neurofeedback as Combined Therapeutic Interventions to Target Glutamatergic Neurotransmission in Alcohol Use Disorder
Brief Title: Ketamine and Neurofeedback as Combined Therapeutic Interventions to Target Glutamatergic Neurotransmission in Alcohol Use Disorder
Acronym: Nektar
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. med. Marcus Herdener (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Marcus Herdener, Principal Investigator, Head of Center for Addictive Disorders, Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-02294
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Abuse/Dependence; Alcohol Use Disorder (AUD); Alcoholism
Keywords: Alcohol Use Disorder; Alcoholism; Alcohol Dependence; Ketamine; Glutamate; Placebo-controlled; Neurofeedback Training; Realtime fMRI; Therapeutic effects; Mechanistic effects
MeSH Terms: conditions — Alcoholism | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Phase II, randomised, placebo-controlled, double blind, parallel group, single centre study investigating ketamine and neurofeedback as combined therapeutic interventions to target glutamatergic neurotransmission in alcohol use disorder.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rt-fMRI NFT / Ketamine (Experimental): Participants get real time neurofeedback based on an experimental regions' activity and receive 0.8 mg ketamine (i.v.) per kilogram bodyweight.
  Interventions: Drug: Ketamine; Behavioral: Real-time fMRI Neurofeedback Training
- sham rt-fMRI NFT / Ketamine (Experimental): Participants get a real time neurofeedback based on a control regions' activity, which serves as a sham region and receive 0.8 mg ketamine (i.v.) per kilogram bodyweight.
  Interventions: Drug: Ketamine; Behavioral: Sham Neurofeedback Training/ Ketamine
- rt-fMRI NFT / Placebo (Experimental): Participants get real time neurofeedback based on an control regions' activity and receive a 0.9% NaCL infusion (placebo).
  Interventions: Behavioral: Real-time fMRI Neurofeedback Training; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — A single dose of ketamine 0.8 mg ketamine (i.v.) per kilogram bodyweight
  Arms: rt-fMRI NFT / Ketamine; sham rt-fMRI NFT / Ketamine
Behavioral: Real-time fMRI Neurofeedback Training — Participants will undergo a closed-loop rt-fMRI paradigm over 25 minutes. Participants will be instructed to use strategies to downregulate cue-induced cravings. The Intensity of cues will adjust based on the participants neural activity in response to cues. This dynamic feedback mechanism allows for personalized training aimed at improving the participant's ability to manage cravings.
  Arms: rt-fMRI NFT / Ketamine; rt-fMRI NFT / Placebo
Drug: Placebo — Single dose of placebo (0.9% NaCl infusion)
  Arms: rt-fMRI NFT / Placebo
Behavioral: Sham Neurofeedback Training/ Ketamine — Participants get a real time neurofeedback based on a control regions' activity, which serves as a sham region and receive 0.8 mg ketamine (i.v.) per kilogram bodyweight. The use of sham-NFT allows for a rigorous assessment of the specific effects of combined rt-fMRI NFT and ketamine by controlling for non-specific factors such as expectancy effects or the therapeutic context.
  Arms: sham rt-fMRI NFT / Ketamine

SUMMARY:
The goal of this clinical trial is to learn about the effects of the combination of ketamine and realtime functional magnetic resonance imaging (fMRI) neurofeedback training on the treatment of individuals with alcohol use disorder (AUD). The main questions the investigators aim to answer are:

* Can the investigators observe a positive, significant therapeutic effect by comparing changes in alcohol use via i) mean alcohol use per day, ii) heavy drinking days one month after the last treatment intervention?
* Are changes in glutamatergic neurotransmission in the nucleus accumbens related to cue-induced cravings in individuals with AUD?
* Is there a significant, ketamine-dependent change in glutamate levels in the nucleus accumbens?

Participants will be given ketamine or placebo and real-time fMRI neurofeedback (rt-fMRI NFT) or sham rt-fMRI NFT.

The investigators will compare three intervention groups to investigate the effects of the stand-alone effects as well as potential synergies between the combination of pharmacological and non-pharmacological intervention.

DETAILED DESCRIPTION:
For decades, addiction research has focused predominantly on the dopaminergic system. However, preclinical research suggests that alterations of glutamatergic neurotransmission within the nucleus accumbens (NAcc) are crucial for cue-induced drug-seeking behavior, at least in animal models of addiction (Kalivas, 2009). In line with this, three randomized controlled trials have been conducted exploring ketamine as a treatment for alcohol use disorder (AUD) or harmful drinking, each combining ketamine with either memory retrieval destabilization procedures or psychological therapy (Dakwar et al., 2020a; Das et al., 2019a; Grabski et al., 2022a). While ketamine consistently reduced alcohol use in these studies, the variability in treatment responses highlights the need for further investigation into the role of the glutamate system in AUD as well as optimal treatment approaches that maximize safety and efficacy for patients.

Given the significant need to advance both mechanistic and clinical understanding of AUD, this study aims to: (1) explore the role of glutamatergic neurotransmission in AUD; (2) determine whether ketamine can modulate potentially pathophysiological altered glutamate neurotransmission, and how such modulation may be influenced by ketamine metabolism ; and (3) optimize ketamine as a treatment for AUD by leveraging synergies between the additional biological mechanism of action of ketamine (i.e., induced neuroplasticity) and a targeted non-pharmacological neuromodulatory intervention, such as neurofeedback training (NFT), to maximize clinical outcomes.

To evaluate both the mechanistic and therapeutic effects of a single ketamine infusion and rt-fMRI NFT as well as their combined application on AUD, we will assess glutamatergic signalling in the NAcc, changes in neuroplasticity via BDNF, inter-individual differences in the metabolism of ketamine, and clinical symptoms in individuals with AUD.

Therefore, in this randomized, placebo-controlled, double blind, parallel group, single centre study we investigate the extend to which a single administration of ketamine and neurofeedback training, as well as the combination of the two interventions can restore neurobiological changes related to alcoholism and what effect this new treatment method has on the symptoms of AUD.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* In- and outpatients aged 18 to 65 years of all sexes.
* DSM-IV diagnosis of alcohol use disorder (mild - severe).
* Motivation to reduce or stop alcohol use
* Normal level of language comprehension (German or Swiss-German)
* Good physical health with no unstable medical conditions
* Participants of childbearing potential must use an effective and established method of contraception for the entire study duration
* Comply with the study protocol as explained by investigator

Exclusion Criteria:

* History of DSM-IV severe drug dependence other than alcohol (except for caffeine or nicotine) and any opiod use disorder within two months prior to enrolment.
* Hallucinogen and ketamine use 3 months prior to study participation (including regular microdosing).
* Alcohol withdrawal symptoms at any of the treatment visits (V2 and V3) (CIWA-Ar Scale >9).
* Current or lifetime psychotic disorders
* History of severe substance-induced psychosis
* Current or lifetime bipolar I or II disorders
* Current suicidality
* Previous suicide attempts during the last 2 years
* High risk of adverse emotional and behavioral reactions
* Unmedicated or unstable hypertension
* Severe illness (e. g. myocardial ischemia or arrythmias, severe pulmonary secretions, glaucoma, congestive heart failure or angina, significant renal or hepatic impairment)
* Acute infection (e. g. pulmonary or upper respiratory tract infection)
* Insufficient treated or uncorrected hyperthyroidism
* Severe central nervous system related traumas or disorders (e. g. stroke, cerebral trauma with loss of consciousness over more than 24h, epilepsy)
* During the study, new use or dose changes of already existing concomitant medication without prior informing the investigators.
* Taking medications that are known to modualte uridine diphosphate glucuronosyltransferase-enzyme
* Medication directly affecting glutamate signaling (e. g. anticonvulsant medication)
* Inhibitors of UGT1A9 and 1A10 should be discontinued at least five half-lives prior to the administration of ketamine.
* Monoamine oxidase and aldehyde or alcohol dehydrogenase inhibitors should be discontinued at least 5 half-lives prior to the dose of ketamine.
* Pregnancy or lactation
* Women of childbearing potential with no use of medically accepted contraceptive (e. g. condoms, contraceptive diaphragm, birth control pill, hormone injection, intrauterine device)
* BMI < 17 or > 35
* Allergy, hypersensitivity, or other adverse reaction to previous use of ketamine
* Contradictions to magnetic resonance imaging
* Concurrent participation in other clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in mean alcohol use per day | Starting immediately after the intervention visit 2 and ending 4 weeks later (integration visit).
  Change in mean alcohol use per day. Alcohol use is measured via a combination of the digital app and the Timeline Follow-Back Questionnaire.
Change in heavy drinking days | Starting immediately after the intervention visit 2 and ending 4 weeks later (integration visit).
  Change in heavy drinking days. Defined as five or more standard units of alcohol in a day for a man and four or more standard units of alcohol in a day for a woman. Alcohol use is measured via a combination of the digital app and the Timeline Follow-Back Questionnaire.

SECONDARY OUTCOMES:
Changes in glutamat levels during craving | During the intervention visit 1a and 1 week later during the intervention visit 2.
  Changes in glutamatergic signalling in the NAcc measured via Magnetic Resonance Spectroscopy (MRS) during craving vs neutral cue exposure.
Changes in Brain Derived Neurotrophic Factor | During the intervention visit 2 at baseline 30 minutes before and 2 hours after infusion start.
  Treatment-induced changes in neuroplasticity assessed using the brain derived neurotrophic factor (BDNF) through blood analysis.
Individual variations in ketamine pharmacokinetics | During the intervention visit 2 at baseline, 45 minutes, 1 hour 30 minutes before, and 2 hours 30 minutes after infusion start.
  Changes in ketamine plasma concentrations and its metabolites measured via blood samples taken.
Predictive value of baseline rs-fMRI for treatment response | Between 1 and 2 weeks after baseline (screening visit) during the intervention visit 1a.
  Predictive value of rs-fMRI for treatment response assessed via the two primary outcomes
Changes in alcohol use in blood alcohol metabolites | At baseline (screening visit) and 4 weeks later (integration visit).
  Blood samples will be collected to analyse markers of alcohol use. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyltransferase (GGT) and Phosphatidyl Ethanol (PEth) will be analysed from blood samples.
Severity of alcohol use disorder | From baseline (screening visit) until 6 months later (follow-up survey II).
  Changes in severity of alcohol use disorder score assessed by the Obsessive Compulsive Drinking Scale, ranging from 0 to 56, where higher scores indicate more compulsive behaviors and obsessive thoughts to use alcohol.
Changes in alcohol abstinence ability | From baseline (screening visit) until 6 months later (follow-up survey II).
  Changes in individuals confidence in their ability to abstain from alcohol in high risk situations assessed with the Alcohol Abstinence Self-Efficacy Scale, ranging from 0 to 160, where higher scores indicate higher self-confidence in the ability to avoid drinking.
Experience of alcohol craving | From baseline (screening visit) until 6 months later (follow-up survey II).
  The Visual Analogue Scale for Alcohol Craving on a scale ranging from 0 to 100, where higher scores indicate higher subjective experience of craving.
Depressive symptoms | From baseline (screening visit) until 6 months later (follow-up survey II).
  Changes in depressive symptoms measured with Beck Depression Inventory. The scale ranges from 0 to 63 where higher scores indicate more severe depressive symptoms.
Experience of pleasure across different domains | From baseline (screening visit) until 6 months later (follow-up survey II).
  Changes in the experience of pleasure across different domains assessed by the Domains of Pleasure Scale, ranging from 0 to 210, where a higher score indicates a higher experience of pleasure.
Hedonic capacity | From baseline (screening visit) until 6 months later (follow-up survey II).
  Changes in hedonic capacity measured by the Trait Hedonic Capacity Scale, ranging from 16 to 80, where a higher score indicates a higher hedonic capacity.
Perceived quality of life | From baseline (screening visit) until 6 months later (follow-up survey II).
  Changes in the perceived quality of life assessed with the Quality of Life Scale, ranging from 0 to 400, whereas higher scores indicate higher perceived quality of life.
Posttraumatic stress symptoms | From baseline (screening visit) until 6 months later (follow-up survey II).
  Changes in posttraumatic stress symptoms measured with Posttraumatic Stress Disorder Checklist for DSM-5. The scale ranges from 0 to 80, where higher scores indicate more severe posttraumatic stress symptoms.
Perceived stress | From baseline (screening visit) until 6 months later (follow-up survey II).
  Changes in perceived stress assessed with a subscale of the Stress & Coping Inventory, ranging from 21 to 147, where higher scores indicate higher perceived stress.
Subjective effects of ketamine infusion | 2 hours after the ketamine infusion (intervention visit 2).
  Assess the acute subjective effects of the infusion with the Five-Dimension Altered State of Consciousness Questionnaire (5D-ASC), ranging from 0 to 100, where higher scores indicate the occurence of altered states of consciousness.
Effects of ketamine infusion on mystic experiences | 2 hours after the ketamine infusion (intervention visit 2).
  Assess the acute subjective effects of the infusion with the Hood's Mysticism Scale, ranging from 20 to 100 where higher scores indicate the occurence of mystic experiences.
Neurofeedback Experience | After neurofeedback training (intervention visit 1b) and up to two weeks later (intervention visit 2).
  The Neurofeedback Post Questionnaire (NF-PostQ) asks participants about their used strategies and experiences during neurofeedback training.
Daily alcohol use and craving | From baseline (screening visit) up to 5 months later (one month prior to follow-up survey II).
  A Digital app (SEMA3) will document daily alcohol craving and alcohol use using an Ecological Momentary Assessment method.
Alcohol use in urine alcohol metabolites | From baseline (screening visit) up to one month later (Integration visit)
  Changes in alcohol metabolites via urine analyses as objective measure of alcohol use.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric University Zurich, University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Our data will be published on the website of Open Science Framework.
Supporting Information: Study Protocol, ICF
Time Frame: After the publication of our data.